CLINICAL TRIAL: NCT01692028
Title: A Novel Approach Localizes the Association of Vitamin D Status With Insulin Resistance to One Region of the 25(OH)D Continuum.
Brief Title: Identification of the Region of Vitamin D Responsiveness
Acronym: GRH-PN01
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: GRH-PN01
Record Dates: First submitted 2012-09-13; First posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes; Hypertension
Keywords: vitamin D; Associational study
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: low vitamin D status is associated with increased insulin resistance and increased blood pressure.

Approach: Multiple regression analysis of information extracted from a large database accumulated by a Canadian health foundation, specifically evaluating statistical associations between serum 25(OH)D levels and insulin responsiveness measures as well as blood pressure, after adjusting these variables for BMI, age, sex, and waist circumference.

DETAILED DESCRIPTION:
Data obtained from the entry records of 4,116 adult men and women in Calgary,Alberta previously enrolled in the Pure North S'Energy Foundation's health program. Individuals with a clinical diagnosis of diabetes mellitus or a HOMA-IR value above 16 were excluded. Standard statistical analyses carried out. An association between 25(OH)D and the endpoints of interest was first established. The residual values after adjusting HOMA-IR, serum insulin, QUICKI, and blood pressure for BMI, age, sex, and waist circumference were then regressed against serum 25(OH)D using 40-percentile data blocks, stepping upward from the lowest 25(OH)D values by 5 percentile increments through the 7th decile. Regression coefficients are then computed for each data block and each outcome variable. The location (along the 25(OF)D continuum) of the largest and most statistically significant coefficients is noted, and regions of null response noted as well.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18

Exclusion Criteria:

* Diabetes
* Elevated HOMA-IR (>16)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults living in or near Calgary and associated with the oil and gas industries
Sampling Method: Non-Probability Sample
Enrollment: 4116 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | Observational/cross-sectional study
  A composite measure of insulin resistance (HOMA-IR)

SECONDARY OUTCOMES:
Blood pressure | cross-sectional study
  Blood Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Pure North S'Energy Foundataion, Calgary, Alberta, Canada